CLINICAL TRIAL: NCT03802162
Title: An Open-label, Randomized, Multiple-dosing Parallel Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-355 With D797 and D324 in Healthy Subjects
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-355
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 179BE18029
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's disease; CKD-355
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CKD-355A (Experimental)
  Interventions: Drug: CKD-355A (D797/Memantine HCl 20mg)
- CKD-355B (Experimental)
  Interventions: Drug: CKD-355B (D797/Memantine HCl 20mg)
- D797, D324 (Active Comparator)
  Interventions: Drug: D797; Drug: D324 (Memantine HCl 10mg)

INTERVENTIONS:
Drug: CKD-355A (D797/Memantine HCl 20mg) — once a day
  Arms: CKD-355A
Drug: CKD-355B (D797/Memantine HCl 20mg) — once a day
  Arms: CKD-355B
Drug: D797 — once a day
  Arms: D797, D324
Drug: D324 (Memantine HCl 10mg) — twice a day
  Arms: D797, D324

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of CKD-355.

DETAILED DESCRIPTION:
An open-label, randomized, multiple-dosing parallel study to evaluate the pharmacokinetics, safety and tolerability of CKD-355 with D797 and D324 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult older than 19 years and less than 55 years at the time of screening
2. BMI 18.5~29.9 kg/m2 and body weight more than 50kg
3. Subjects who have consented to the use of appropriate double- pregnancy contraceptive methods up to two months after the last investigational product and not to provide sperm for men
4. Subjects who sign on an informed consent form willingly

Exclusion Criteria:

1. Subjects who have a clinically significant disease such as respiratory, hepatic, kidneys, blood, gastrointestinal, endocrine, immune system, skin, nercous and mental disease.
2. Subjects who have acute disease within 28 days prior to the first administration
3. Subjects who have history that may affect the ADME
4. Subjects who have clinically significant chronic disease
5. Women who are nursing, pregnant or positive on pregnancy test
6. Subjects who have clinically significant allergic diseases
7. Subjects with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
8. Subjects who are known to be hypersensitive to the drug or its components
9. Subjects who have been found to be positive in serological tests (HBs antigen, HCV antibody and HIV antibody)
10. Subjects with creatinine clearance <60 ml / min
11. Subjects whose AST or ALT levels exceeded 2.5 times of upper limit of normal range
12. Subjects who taked ETC(Ethical Drug), oriental medicine within 2 weeks and OTC(Over-the-counter Drug), vitamin within 1 week prior to the first administration
13. Subjects who can not eat standard meals provided by the institution.
14. Subjects who donated whole blood within 60 days, donated the components within 20 days or received blood within 30 days
15. Subjects who taked medication for the induction and inhibition of metabolizing enzymes such as barbiturate drugs within 30 days before the first administration
16. Subjects who have had abnormal diets that can affect the ADME of the drug within 30 days before the first administration (eg, ingestion of grapefruit juice>1 L / day)
17. Subjects who participate in the other clinical trial within 90 days prior to the first administration
18. Subjects who have a history of regular alcohol(alcohol>210g/week) or caffeine(caffeine>5 cups/day)
19. Subjects who smokes more than 10 cigarettes per day within 3 months or cannot discontinue smoking during the clinical trial
20. Subjects who is determined unsuitable to participate in this clinical trial by the investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Cmax of D324 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Max Concentration of D324
AUCt of D324 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Area under the curve of D324
Cmax of D797 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Max Concentration of D797
AUCt of D797 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Area under the curve of D797

SECONDARY OUTCOMES:
Cmin of D324 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Min Concentration of D324
Cmin of D797 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Min Concentration of D797
Tmax of D324 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Time of Max concentration of D324
Tmax of D797 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Time of Max concentration of D797
t½ of D324 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Half-life time of D324
t½ of D797 | 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours
  Half-life time of D797

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea